CLINICAL TRIAL: NCT00376883
Title: The Effect of i.v. Bisphosphonate on Health-Related Quality of Life and Skeletal Morbidity for Newly Diagnosed Treatment Demanding Multiple Myeloma. A Prospective Randomised Double Blinded Dose-Effective Study With Cost-Utility Analysis.
Brief Title: Pamidronate Prophylaxis in Multiple Myeloma 30 mg/Month Versus 90 mg/Month
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nordic Myeloma Study Group (Other)
Collaborators: Nordic Cancer Union (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NMSG 08/00; NCU D3-98
Record Dates: First submitted 2006-09-14; First posted 2006-09-15 (Estimated); Last update posted 2007-01-04 (Estimated); Status verified 2007-01

CONDITIONS: Multiple Myeloma
Keywords: multiple myeloma; pamidronate prophylaxis; dose comparison; quality of life; skeletal event; response; survival
MeSH Terms: conditions — Multiple Myeloma | interventions — Pamidronate

INTERVENTIONS:
Drug: pamidronate

SUMMARY:
Multiple myeloma is a malignant hematological disease dominated by monoclonal plasma cells in the bone marrow. Major symptoms are related to the bones due to an increased bone resorption and a decreased bone formation leading to bone pain and increased risk of fractures. The normal osteoclasts are responsible for bone degradation through stimulation from the malignant plasma cells. Bisphosphonates have been shown to inhibit the osteoclast activity but may have serious side-effects due to renal toxicity and the optimal dose have not been established.

In a randomized double blinded design it is aim to compare the standard of monthly injections of 90 mg pamidronate with 30 mg.

The primary end-point is physical function estimated by EORTC QLQ-C30 questionnaire at 12 months after starting the treatment in newly diagnosed treatment demanding multiple myeloma. Secondary end-points are skeletal related events, cost-utility analysis, response, response duration and survival and quality of life with respect to fatigue and pain.

DETAILED DESCRIPTION:
Patients with newly diagnosed treatment demanding multiple myeloma are after informed consent and approved inclusion criteria randomised by telephone call to Copenhagen Trial Unit (CTU) and information on the target dose is send to the distributor, Amgros, and the local pharmacy for preparation of the pamidronate solution. Infusion is given for 2½ hours.

Before starting treatment the patient has to fulfil the first EORTC QLQ-C30 questionnaire that is send to the quality of life secretariat in Oslo, Norway. Subsequent questionnaires are mailed directly to the patients every third month.

The infusions are continued for 3 years and may be extended further upon the patient's request.

Every third month the number of skeletal event, the response and complications are recorded.

Skeletal X-rays are performed 9 and 24 months after starting the treatment.

ELIGIBILITY:
Inclusion Criteria:

* New diagnosed multiple myeloma with treatment demanding disease

Exclusion Criteria:

* Life-expectancy less than 3 months, another active malignant disease, treatment with bisphosphonates for more than 3 months within the last 6 months, patients with creatinine above 400 µmol/l 4 weeks after starting chemotherapy, patients who cannot cooperate for monthly infusions, patients who do not give their informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500
Dates: Start 2000-01; Study Completion 2006-10

PRIMARY OUTCOMES:
Physical function at 12 months estimated by EORTC QLQ-C30 questionnaire

SECONDARY OUTCOMES:
Skeletal related event (time to first SRE)
Cost-utility analysis
Subgroup analysis (conventional chemotherapy vs. high dose chemotherapy with stem cell support)
Response, recons duration, survival
Quality of Life estimated by fatigue and pain according to EORTC QLQ-C30

CONTACTS AND LOCATIONS:
Overall Officials: Peter Gimsing, Ass. prof., Principal Investigator — Nordic Myeloma Study Group
Locations (14):
- Denmark (4):
  - Department of Haematology B, Aalborg Hospital, University of Aarhus, Aalborg
  - Hæmatologisk afd., Århus Universitetshospital, Aarhus
  - Department of Haematology, Herlev University Hospital, Herlev
  - Department of Hematology L, Rigshospitalet, København Ø
- Norway (4):
  - Hematologisk seksjon, med avd, Haukeland Universitetssykehus, Bergen
  - Hematologisk avdeling Ullevål Sykehus, Oslo
  - Med avd B, Hematologisk seksjon, Universitetssykehuset Nord Norge, Tromsø
  - Hematologisk seksjon, St.Olav Hospital, Trondheim
- Sweden (6):
  - Sahlgrenska Universitetsjukhuset Östra, Gothenburg
  - Hematologkliniken, Universitetssjukhuset, Linköping
  - Medicinklin, Universitetssjukhuset MAS,, Malmo
  - Medicinkliniken, Universitetssjukhuset, Örebro
  - Medicinklin, sekt för hematologi, Norrlands Universitetssjukhus, Umeå
  - Medicinklinikken Akademiska sjukhuset, Uppsala

REFERENCES:
- [Derived] Gimsing P, Carlson K, Turesson I, Fayers P, Waage A, Vangsted A, Mylin A, Gluud C, Juliusson G, Gregersen H, Hjorth-Hansen H, Nesthus I, Dahl IM, Westin J, Nielsen JL, Knudsen LM, Ahlberg L, Hjorth M, Abildgaard N, Andersen NF, Linder O, Wisloff F. Effect of pamidronate 30 mg versus 90 mg on physical function in patients with newly diagnosed multiple myeloma (Nordic Myeloma Study Group): a double-blind, randomised controlled trial. Lancet Oncol. 2010 Oct;11(10):973-82. doi: 10.1016/S1470-2045(10)70198-4. PMID 20863761